CLINICAL TRIAL: NCT00465933
Title: Treatment of Acute Promyelocytic Leukemia: Remission Induction With ATRA + Idarubicin (AIDA) Risk Adapted Intensity of Consolidation and Addition of ATRA Maintenance With ATRA + Methotrexate + Mercaptopurine Salvage Therapy for Molecular and Haematological Relapses
Brief Title: Treatment of Acute Promyelocytic Leukemia With All-Trans Retinoic Acid (ATRA) and Idarubicin (AIDA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pethema LPA-99 protocol
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute Promyelocytic Leukemia; AIDA
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

INTERVENTIONS:
Drug: AIDA

SUMMARY:
The purpose of this study is to evaluate the efficacy of all-trans retinoic acid (ATRA) and idarubicin (AIDA) with a dose reduction in patients older than 70 years of age in the remission induction of acute promyelocytic leukemia (APL).

With regard to the induction, the excellent results obtained by the combination of ATRA and idarubicin (AIDA), especially in terms of antileukemic efficacy (1% of resistance), do not support the introduction of substantial changes in this combination. However, given that most of the induction failures were caused by complications, especially of a hemorrhagic nature, and that these had a major impact in the hyperleukocytic forms and in patients older than 70 years of age, the induction was modified as follows:

1. Reduction of idarubicin dose in patients older than 70 years of age (three days instead of four);
2. Early administration of corticosteroid therapy in all patients as ATRA syndrome prophylaxis. A preliminary analysis of the Italian Group for Adult Hematologic Diseases (Gruppo Italiano Malattie Ematologiche dell'Adulto, GIMEMA) has shown that low dose prednisone use in a prophylactic manner appears to reduce the incidence and severity of the ATRA syndrome, which could also have a favorable impact on the hemorrhagic mortality (non-published data); and
3. Treatment of the hyperfibrinolysis with an antifibrinolytic agent (tranexamic acid). It has been recently reported that APL cells present abnormally high levels of annexins (especially annexin II), and that these levels may provide the fundamental mechanism for the hemorrhagic complications in APL by increasing the production of t-PA dependent plasmin. These findings provide new reasons for the introduction of tranexamic acid in the hemorrhagic prophylaxis of APL.

DETAILED DESCRIPTION:
Induction chemotherapy:

All-trans retinoic acid, will be administered by mouth (PO) from the first day at a dose of 45 mg/m²/day, fractionated into 2 doses.

In patients aged < 20 years, the ATRA dose will be reduced to 25 mg/m²/day fractionated into 2 doses.

The treatment with ATRA will continue until a CR is achieved or for a maximum of 90 days in the case of persistence of atypical promyelocytes in the bone marrow.

Idarubicin, 12 mg/m² on days 2, 4, 6 and 8 of treatment by slow intravenous infusion (20 minutes).

In patients older than 70 years of age only 3 doses of idarubicin will be given on days 2, 4, and 6.

Supporting measures:

Prednisone, 0.5 mg/kg/day days 1 to 15. Tranexamic acid, 100 mg/kg/day in continuous perfusion, if platelets < 50 x 10^9/L or evident clinical-biological signs of coagulopathy. This treatment will be discontinued if the platelet counts are > 50 x 10^9/L.

Transfusion of platelet concentrates to keep up counts above 30 x 10^9/L during the first 10 days and PRC to maintain hemoglobin levels greater than 9 g/dL.

Prophylactic heparin should not be used.

ELIGIBILITY:
Inclusion Criteria:

* Age <= 75 years
* ECOG = 3.
* Morphological diagnosis of M3 or M3v. Those cases without typical morphology but with PML-RARa rearrangement may also be included.
* Genetic diagnosis: t(15;17), PML-RARa rearrangement, monoclonal anti-PML positive. Obviously, the result of these tests may become available after having initiated the treatment based on a tentative morphological diagnosis. The presence of secondary cytogenetic changes associated with t(15;17) is not a reason for exclusion nor do they require a different therapeutic approach.

Exclusion Criteria:

* Age > 75 years (the treatment with this protocol can be considered on an individual basis but these patients will be analysed separately)
* Absence of PML-RARa rearrangement.
* Prior antileukemic chemotherapy.
* Presence of an associated neoplasm.
* Presence of a severe psychiatric disease.
* HIV seropositivity.
* Contraindication for intensive chemotherapy, especially to anthracyclines.
* Serum creatinine = 2.5 mg/dL.
* Bilirubin, alkaline phosphatase, or SGOT > 3 times the upper normal limit
* Positive pregnancy test.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-03; Primary Completion 2007-08 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of AIDA with a dose reduction in patients older than 70 years of age in the remission induction of APL | 6 months
To evaluate the impact on morbidity and mortality of the prophylactic measures included in induction therapy (low dose prednisone and tranexamic acid) | 1 year
To evaluate the toxicity of the induction, consolidation, and maintenance chemotherapy | 2 years
To evaluate the impact on the event free survival, disease free survival and global survival in each relapse risk group | 5 years
To evaluate the rates of molecular remission (PML/RARa negative by RT-PCR) in the successive therapeutic phases with special emphasis on patients with a higher risk for relapse | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sanz Miguel Angel, Dr, Study Chair — Hospital La Fe de Valencia
Locations (2):
- Spain (2):
  - Hospital La Fe de Valencia, Valencia, Valencia
  - Basurtuko Ospitalea, Basurto

REFERENCES:
- [Background] Miller WH Jr, Kakizuka A, Frankel SR, Warrell RP Jr, DeBlasio A, Levine K, Evans RM, Dmitrovsky E. Reverse transcription polymerase chain reaction for the rearranged retinoic acid receptor alpha clarifies diagnosis and detects minimal residual disease in acute promyelocytic leukemia. Proc Natl Acad Sci U S A. 1992 Apr 1;89(7):2694-8. doi: 10.1073/pnas.89.7.2694. PMID 1372989
- [Background] Slack JL: Recent advances in the biology and treatment of acute promyelocytic leukemia. Educational Book of the 34th Meeting of the American Society of Clinical Oncology, Los Angeles, CA 1998, p.54-65
- [Background] Mandelli F, Diverio D, Avvisati G, Luciano A, Barbui T, Bernasconi C, Broccia G, Cerri R, Falda M, Fioritoni G, Leoni F, Liso V, Petti MC, Rodeghiero F, Saglio G, Vegna ML, Visani G, Jehn U, Willemze R, Muus P, Pelicci PG, Biondi A, Lo Coco F. Molecular remission in PML/RAR alpha-positive acute promyelocytic leukemia by combined all-trans retinoic acid and idarubicin (AIDA) therapy. Gruppo Italiano-Malattie Ematologiche Maligne dell'Adulto and Associazione Italiana di Ematologia ed Oncologia Pediatrica Cooperative Groups. Blood. 1997 Aug 1;90(3):1014-21. PMID 9242531
- [Background] Fenaux P, Chastang C, Chevret S, Sanz M, Dombret H, Archimbaud E, Fey M, Rayon C, Huguet F, Sotto JJ, Gardin C, Makhoul PC, Travade P, Solary E, Fegueux N, Bordessoule D, Miguel JS, Link H, Desablens B, Stamatoullas A, Deconinck E, Maloisel F, Castaigne S, Preudhomme C, Degos L. A randomized comparison of all transretinoic acid (ATRA) followed by chemotherapy and ATRA plus chemotherapy and the role of maintenance therapy in newly diagnosed acute promyelocytic leukemia. The European APL Group. Blood. 1999 Aug 15;94(4):1192-200. PMID 10438706
- [Background] Frankel SR, Eardley A, Heller G, Berman E, Miller WH Jr, Dmitrovsky E, Warrell RP Jr. All-trans retinoic acid for acute promyelocytic leukemia. Results of the New York Study. Ann Intern Med. 1994 Feb 15;120(4):278-86. doi: 10.7326/0003-4819-120-4-199402150-00004. PMID 8291820
- [Background] Burnett AK, Grimwade D, Solomon E, Wheatley K, Goldstone AH. Presenting white blood cell count and kinetics of molecular remission predict prognosis in acute promyelocytic leukemia treated with all-trans retinoic acid: result of the Randomized MRC Trial. Blood. 1999 Jun 15;93(12):4131-43. PMID 10361110
- [Background] Tallman MS, Andersen JW, Schiffer CA, Appelbaum FR, Feusner JH, Ogden A, Shepherd L, Willman C, Bloomfield CD, Rowe JM, Wiernik PH. All-trans-retinoic acid in acute promyelocytic leukemia. N Engl J Med. 1997 Oct 9;337(15):1021-8. doi: 10.1056/NEJM199710093371501. PMID 9321529
- [Background] Asou N, Adachi K, Tamura J, Kanamaru A, Kageyama S, Hiraoka A, Omoto E, Akiyama H, Tsubaki K, Saito K, Kuriyama K, Oh H, Kitano K, Miyawaki S, Takeyama K, Yamada O, Nishikawa K, Takahashi M, Matsuda S, Ohtake S, Suzushima H, Emi N, Ohno R. Analysis of prognostic factors in newly diagnosed acute promyelocytic leukemia treated with all-trans retinoic acid and chemotherapy. Japan Adult Leukemia Study Group. J Clin Oncol. 1998 Jan;16(1):78-85. doi: 10.1200/JCO.1998.16.1.78. PMID 9440726
- [Background] Head D, Kopecky KJ, Weick J, Files JC, Ryan D, Foucar K, Montiel M, Bickers J, Fishleder A, Miller M, et al. Effect of aggressive daunomycin therapy on survival in acute promyelocytic leukemia. Blood. 1995 Sep 1;86(5):1717-28. PMID 7655004
- [Background] Bernard J, Weil M, Boiron M, Jacquillat C, Flandrin G, Gemon MF. Acute promyelocytic leukemia: results of treatment by daunorubicin. Blood. 1973 Apr;41(4):489-96. No abstract available. PMID 4510926
- [Background] Sanz MA, Jarque I, Martin G, Lorenzo I, Martinez J, Rafecas J, Pastor E, Sayas MJ, Sanz G, Gomis F. Acute promyelocytic leukemia. Therapy results and prognostic factors. Cancer. 1988 Jan 1;61(1):7-13. doi: 10.1002/1097-0142(19880101)61:13.0.co;2-6. PMID 3422032
- [Background] Petti MC, Avvisati G, Amadori S, Baccarani M, Guarini AR, Papa G, Rosti GA, Tura S, Mandelli F. Acute promyelocytic leukemia: clinical aspects and results of treatment in 62 patients. Haematologica. 1987 Mar-Apr;72(2):151-5. No abstract available. PMID 3114070
- [Background] Marty M, Ganem G, Fischer J, Flandrin G, Berger R, Schaison G, Degos L, Boiron M. [Acute promyelocytic leukemia: retrospective study of 119 patients treated with daunorubicin]. Nouv Rev Fr Hematol (1978). 1984;26(6):371-8. French. PMID 6597407
- [Background] Avvisati G, Mandelli F, Petti MC, Vegna ML, Spadea A, Liso V, Specchia G, Bernasconi C, Alessandrino EP, Piatti C, et al. Idarubicin (4-demethoxydaunorubicin) as single agent for remission induction of previously untreated acute promyelocytic leukemia: a pilot study of the Italian cooperative group GIMEMA. Eur J Haematol. 1990 Apr;44(4):257-60. doi: 10.1111/j.1600-0609.1990.tb00389.x. PMID 2188854
- See also: Spanish Association of Haematology — http://www.aehh.org